CLINICAL TRIAL: NCT02191995
Title: Yoga in the Treatment of Eating Disorders: a Randomized Trial
Acronym: TEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1405S51026
Record Dates: First submitted 2014-05-07; First posted 2014-07-16 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- body awareness yoga (Experimental): body awareness yoga session prior to breakfast meal
  Interventions: Behavioral: yoga
- Control Arm (No Intervention): No intervention

INTERVENTIONS:
Behavioral: yoga
  Arms: body awareness yoga

SUMMARY:
Yoga facilitates the treatment of eating disorders by decreasing symptom severity over time.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the Anna Westin House treatment facility of the Emily Program in MN during timeframe study is being run

Exclusion Criteria:

* declines participation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Participants' level of mood and anxiety | Week 4
  The Positive And Negative Affect Scale will be administered daily prior to and after supper in order to assess anxiety and mood.

SECONDARY OUTCOMES:
Level of eating disorder symptoms | Week 4
  The Eating Disorder Examination-Questionnaire will be administered to evaluate clients' eating disorder symptoms and prevalence.
Participants' ability to tolerance distress | Week 4
  The Distress Tolerance Scale will be administered to follow clients' ability to cope with highly charged emotions.

CONTACTS AND LOCATIONS:
Overall Officials: Dianne Neumark-Sztainer, PhD MPH RD, Principal Investigator — University of Minnesota; Carol Peterson, PhD LP, Principal Investigator — University of Minnesota; Scott Crow, MD, Principal Investigator — University of Minnesota; Lisa Diers, RD LD RYT, Principal Investigator — The Emily Program
Locations (1):
- The Emily Program, Saint Paul, Minnesota, United States